CLINICAL TRIAL: NCT00208117
Title: A Randomized Controlled Trial of Inflammatory Markers, Depressive Symptoms, and Heart Disease
Brief Title: A Trial of Inflammatory Markers, Depressive Symptoms, and Heart Disease
Acronym: CHIME
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unable to enroll subjects
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4976 (Davidson)
Record Dates: First submitted 2005-09-15; First posted 2005-09-21 (Estimated); Last update posted 2012-05-31 (Estimated); Status verified 2012-05

CONDITIONS: Depression; Coronary Artery Disease (CAD); Acute Coronary Syndrome (ACS)
Keywords: depression; inflammation; heart disease; randomized clinical trial; sertraline; simvastatin; placebo
MeSH Terms: conditions — Depression; Coronary Artery Disease; Acute Coronary Syndrome; Inflammation; Heart Diseases | interventions — Sertraline; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Patients randomized to sertraline will receive 50 mg/d for the first 6 weeks. Based on clinical response and tolerability, the dosage will be increased to 2 tablets (100 mg/d) at the end of week 6 until the end of the study (8 weeks). If AEs occur, the dosage will be reduced by 50 mg (1 tablet) at a time, as long as a minimum daily dose of 50 mg is maintained. The psychiatry fellow will be responsible for drug administration and will see all patients weekly. All randomized patients will also be seen at the mid-treatment, post-treatment, and follow-up visits by the study psychiatrist to determine depression symptom severity (HAM-D), assess medical tolerance to the study medications, and ensure patient psychiatric safety. The study psychiatrist will be blinded to treatment allocation.
  Interventions: Drug: Sertraline (Zoloft)
- 2 (Placebo Comparator): To ensure blinding of research assessments and the patient, all medications, including the placebo, will be reformulated into a matching number of identical-appearing pills. All randomized patients will also be seen at the mid-treatment, post-treatment, and follow-up visits by the study psychiatrist to determine depression symptom severity (HAM-D), assess the medical tolerance to the study medications (including placebo), and ensure patient psychiatric safety. The study psychiatrist will be blinded to treatment allocation.
  Interventions: Drug: Simvastatin (Zocor)

INTERVENTIONS:
Drug: Sertraline (Zoloft) — Patients randomized to sertraline will receive 50 mg/d for the first 6 weeks. Based on clinical response and tolerability, the dosage will be increased to 2 tablets (100 mg/d) at the end of week 6 until the end of the study (8 weeks). If adverse events occur, the dosage will be reduced by 50 mg (1 tablet) at a time, as long as a minimum daily dose of 50 mg is maintained.
  Arms: 1
Drug: Simvastatin (Zocor) — The placebo drug will be administered for 8 weeks. To ensure blinding of research assessments and the patient, all medications, including the placebo, will be reformulated into a matching number of identical-appearing pills.
  Arms: 2

SUMMARY:
The purpose of this study is to examine the relationship between depressive symptoms and markers of inflammation, two predictors of heart disease.

DETAILED DESCRIPTION:
Depressive symptoms and inflammatory markers have both been proposed as measures that indicate/precede coronary artery disease (CAD). However, no controlled research study has tested the impact of these two candidate CAD risk factors within the same design to see the directionality of their influence. This study will explore if simvastatin reduces depressive symptoms and if sertraline reduces C-Reactive protein (CRP). Additionally, the recruitment process will help determine the feasibility of a larger trial, powered for significance testing. Three hundred and seventy-five participants will be consented and screened for this study. We expect forty-two otherwise healthy outpatients to have both elevated symptoms and high CRP levels, and be willing to be randomly assigned to sertraline, an antidepressant, simvastatin, a drug with anti-inflammatory properties, or a placebo for 8 weeks. Depressive symptoms and inflammatory indicators will be assessed before treatment (screening and baseline), mid-treatment (after 4 weeks), post-treatment (after 8 weeks), and a follow-up visit (after 12 weeks), using blood tests and depression interviews. We expect that both inflammation and depressive symptoms may be reduced by both medications, but the number of subjects needed to test this hypothesis is not yet known. Hence, this pilot study will be conducted. Knowledge about the inter-dependency of these two CAD risk factors allows the most promising future observational/intervention studies to be designed and conducted.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 60
2. Mild depression
3. Inflammatory markers: CRP > 2

Exclusion Criteria:

1. Non-English or Non-Spanish speakers
2. Active suicidal or homicidal ideation
3. Current alcohol or other substance abuse
4. Psychotic features
5. Current personality disorder
6. History of bipolar depressive disorder
7. Any current psychotic disorder
8. Current major depressive disorder
9. Current depression treatment or treatment within preceding 6 weeks
10. History of chronic liver and/or renal disease
11. Current use or contraindication to any of the tested medications
12. Absence of a response to a previous adequate trial of any of the tested medications
13. Pregnant or lactating women
14. History of coronary artery disease
15. Current use of statins
16. Current, regular aspirin use
17. Antibiotic use within the previous four weeks
18. History of diabetes
19. Inflammatory diseases
20. Meets NCEP guidelines for cholesterol lowering therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2005-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Score on Beck Depression Inventory and C-Reactive Protein Level at weeks 4, 8, and 12 | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Karina W Davidson, PhD, Principal Investigator — Columbia University: Behavioral Cardiovascular Health and Hypertension Program
Locations (1):
- Columbia University Department of General Medicine, New York, New York, United States